CLINICAL TRIAL: NCT02293733
Title: Retrospective Multicenter Observational Study in NSCLC Patients With Epidermal Growth Factor Receptor (EGFR) Activating Mutation Treated First Line by Tyrosine Kinase Inhibitor (TKI)
Brief Title: Retrospective Study in Non Small Cell Lung Cancer (NSCLC) With Epidermal Growth Factor Receptor (EGFR)
Acronym: EGFR-RETRO
Status: Completed | Type: Observational
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Other Study IDs: GFPC 04-2013
Record Dates: First submitted 2014-07-15; First posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: NSCLC Non Small Cells Lung Cancer
Keywords: Retrospective; EGFR; mutation; TKI; NSCLC

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients NSCLC EGFR mutated: This is an observational study, there is no intervention.

SUMMARY:
The purpose of our retrospective study is to describe which circumstances EGFR TKI is continued despite progression according to the usual Response Evaluation CrIteria in Solid Tumours (RECIST) in patients with EGFR activating mutations and acquired resistance to EGFR TKI .We will collect their social and demographic data (age, sex), first Progression Free Survival ( PFS) - from start of EGFR TKI to 1st progression PFS 1- and - from first progression according to RECIST to second progression : PFS2- , Overall Survival (OS) - from diagnosis OS 1 and from first progression OS 2 -, mutational status. We will analyze more closely the mode of progression (site), the therapeutic approach at disease progression. We will define two subgroups: those for whom EGFR TKI was continued at least three months despite progression defined according to RECIST criteria, and those for whom a second-line treatment (chemotherapy without EGFR TKI) was chosen at disease progression. It will be individualized the subgroup of patients in whom it was continued TKI after progression.

DETAILED DESCRIPTION:
Background :

• Lung cancer represents the leading cause of death by cancer in France. Significant advances have been made in recent years on knowledge of oncogenesis of NSCLC in particularly the discovery of specific oncogenic drivers playing major role in oncogenic addiction responsible for the occurrence of NSCLC. Activating mutations of the gene encoding the receptor tyrosine kinase EGFR appeared in a subgroup of patients with NSCLC. In 2010, the search for EGFR mutations in patients with lung cancer was performed in 16,834 patients and the mutation rate was 10.5%. The use of specific inhibitors of EGFR tyrosine kinase in patients with activating mutations of EGFR have shown a significant clinical benefit with a response rate more than 70 % ,with PFS ranging from 9 to 13,1 months and median overall survival from 20 to 30 months. Despite these very good results, all patients develop a resistance to EGFR TKI. This progression is usually defined according to RECIST criteria.

These RECIST criteria were established primarily on studies conducted in patients treated with conventional chemotherapy with few or no targeted therapies. In addition, the mode of action of TKI (blocking signalling pathways involved in cell proliferation, angiogenesis, apoptosis, metastasis ..) is very different from the mode of cytotoxic action (action during cell division). Thus, the use of RECIST does not seem to be the most appropriate way to evaluate the response in patients treated by TKI.

Despite this, the RECIST criteria have been used to demonstrate superiority of EGFR TKI compared to chemotherapy in patients with EGFR activating mutations in first line setting.

In 2010, Pr Jackman proposed a clinical definition of acquired resistance to EGFR TKI :

1. Treatment with a single agent EGFR TKI,
2. Presence of EGFR activating mutation, clinical benefit from treatment with an EGFR TKI
3. Systemic progression of disease according to RECIST or WHO criteria while on continuous treatment with EGFR TKI within the last 30 days TKI
4. No intervening systemic therapy between cessation of EGFR TKI and initiation of new therapy.

Tony Mok , in the accompanying editorial, made some criticism to this definition. He argued that it was not uncommon to find new small slow growing tumor nodules after the dramatic initial response to EGFR TKIs. He stated that in this situation, EGFR TKIs could be continued with benefit for the patients.

Since then, others clinical situations have been described, such as the emergence of one or even more new metastasis located in one single organ (like the brain or bones), which can be controlled by a loco-regional treatment. The authors found that the continuation of EGFR TKIs in these cases allowed control of the disease for a considerable length of time.

More recently, it has been suggested that even loco-regional treatment was not mandatory for EGFR TKIs continuation.

Pr Nishino studied retrospectively 56 patients with EGFR activating mutations and acquired resistance. 88% of patients continued EGFR TKI treatment for at least 2 months beyond progressive disease defined according to RECIST criteria. The median time from RECIST progressive disease to termination of TKI for these patients was 10.1 months (range 2.2 to 64.2 months) and the median overall survival was 31.8 months, which is a rather good result.

Pr Oxnard, in a similar study, found that in 45% of 42 patients with acquired resistance to EGFR TKI, alternate systemic therapy could be delayed for three months or more. These 19 patients had more frequently the exon 19 deletion and were free of cancer related symptoms at RECIST progressive disease.

Another recently published retrospective Japanese study suggested that continuous use of EGFR-TKI beyond progressive disease may prolong overall survival compared with switching to cytotoxic chemotherapy in patients with EGFR activating mutations.

A prospective ASIAN phase II study (ASPIRATION) has been recently completed. It compared the continuous use of erlotinib versus stopping erlotinib at progression according to RECIST criteria. Patients could continue erlotinib if progression was slow (> 6 months stability), asymptomatic minimal increase and/or new cerebral metastasis controlled locally. The patients switch to another systemic treatment if they had rapid progressive disease, extra brain symptomatic metastasis, deterioration of Performance Status (PS) or life threatening complications. The results of this study should be available in December 2014.

Purpose :

The purpose of our retrospective study is to describe which circumstances EGFR TKI is continued despite progression according to the usual RECIST criteria in patients with EGFR activating mutations and acquired resistance to EGFR TKI. This study concerns patients who have began a TKI treatment in first line from 1st JANUARY 2010 to 1st JUNE 2012.We'll collect their social and demographic data (age, sex), first PFS (from start of EGFR TKI: PFS 1) and second (from first progression according to RECIST 1.1 to second progression : PFS2) , OS (from diagnosis OS 1 and from first progression OS2), mutational status, and we will analyze more closely the mode of progression (site), the therapeutic approach at disease progression. We will define two subgroups: those for whom EGFR TKI was continued at least three months despite progression defined according to RECIST criteria, and those for whom a second-line treatment (chemotherapy without EGFR TKI) was chosen at disease progression. It will be individualized the subgroup of patients in whom it was continued TKI after progression.

In this subgroup, it will be searched for a correlation between delaying systemic therapy (second line) by pursuing a EGFR TKI at least 3 months and various parameters:

* Type of EGFR mutation
* Symptoms at disease progression
* Clinical characteristic
* Emergence of new metastases vs increasing size of known targets
* Speed of decay and tumour progression (% per month)
* Delivery of loco-regional treatment when relapse occurs in a single site
* PFS (PFS1 and PFS2) and OS (OS1) from the first progression in this group will be compared to the general population (population for which there was TKI stop to the progression) with EGFR activating mutations.

ELIGIBILITY:
Eligibility criteria:

* Inclusion criteria:

  * NSCLC patients with activating mutations of EGFR
  * First-line treatment with a TKI monotherapy
  * Measurable lesion according to RECIST 1.1
  * Age> 18 years
  * secondary or acquired resistance of EGFR TKIs according to the jackman criteria
  * patients for whom it was started a TKI treatment in first line from January 2010 until June 2012 (patients who received 1 Chemotherapy cycle could be included).
* Exclusion criteria:

  * Patients with small cell carcinoma
  * Patients without EGFR mutation
  * Patients not treated with EGFR TKI in first line treatment
  * Not measurable lesion to RECIST 1.1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC with activating mutations of EGFR and who began a treatment by TKI in first line from 1st January 2010 to 1st June 2012.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients continuing TKI at 1st progression and proportion of patients discontinuing EGFR TKI at 1st progression. Analysis of the therapeutic management in the 2 groups. This outcome consists in multiple measures. | Patients are followed up to 48 Months maximum
  • Primary outcome: the therapeutic management of secondary resistance to EGFR TKI (erlotinib or gefitinib) in patients with advanced NSCLC with EGFR activating mutation. Comparison of demographic, clinical, biological features and outcome of patients continuing EGFR TKI at progression versus interrupting TKI at progression. Composite measures will be performed : demographic and clinical data, Progression Free Survival (PFS), Overall Survival (OS), mutational status, mode of progression, therapeutic approach at progressive disease in patients with EGFR mutation treated in first line by EGFR TKI (all population and subgroups : patients receiving EGFR-TKI at progressive disease - Group 1 -, patients discontinuing EGFR TKI at progressive disease - Group 2- ).

SECONDARY OUTCOMES:
Comparison of clinical data and outcome of patients | Patients are followed up to 48 Months maximum
  A comparison of clinical data and outcome of patients receiving EGFR-TKI beyond progressive disease (group 1) versus discontinuing EGFR-TKI at progressive disease (group 2) will be made.
Median Progression Free Survival (PFS) | Patients are followed up to 48 Months maximum
  • Median Progression Free Survival (PFS) (months) in group 1 and 2 - from start of EGFR TKI to first progression : PFS 1- and - from first progression to second progression : PFS2 -.
Univariate and multivariate analysis of Median over survival (OS) | Patients are followed up to 48 Months maximum
  • Univariate an multivariate analysis of OS between the 2 groups will be adjusted using the Cox model. Variables as : age, gender, PS, histology, brain metastasis, EGFR mutations (deletions in exon 19, L858R mutations), TKI continued or TKI stopped at progression, metastasis number and site, will be considered for adjustment.
Univariate and multivariate analysis of OS | Patients are followed up to 48 Months maximum
  • Univariate and multivariate analysis of OS between the 2 groups will be adjusted using the Cox model. Following variables will be considered for adjustment: age, gender, PS, histology, brain metastases, EGFR mutations (deletions in exon 19, L858R mutations), TKI continued to progression or TKI stopped at progression, metastasis number and site

CONTACTS AND LOCATIONS:
Overall Officials: AULIAC JA Jean-Bernard, MD, Principal Investigator — Hôpital F. Quesnay 2 bd de Sully 78201 MANTES LA JOLIE; GERVAIS RG Radj, MD, Study Director — Centre François Baclesse 3 avenue du Général Harris 14076 CAEN CEDEX 05
Locations (24):
- France (24):
  - Centre Hospitalier D Argenteuil, Argenteuil, Val D'oise
  - Site 12, Aix-en-Provence
  - Centre Hospitalier Universitaire, Angers
  - Centre Hospitalier du Morvan, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier René Dubos, Cergy-Pontoise
  - Site 33, Créteil
  - Site 07, Draguignan
  - Site 32, Elbeuf
  - Site 04, Gap
  - Centre Hospitalier Les Oudairies, La Roche-sur-Yon
  - Hospital du Cluzeau, Limoges
  - Site 00, Limoges
  - Centre Hospitalier Régional, Longjumeau
  - Site 25, Mantes-la-Jolie
  - Site 06, Marseille
  - Site 01, Meaux
  - Site 19, Périgueux
  - Site 20, Rennes
  - Site 18, Rouen
  - Site 17, Rouen
  - Hôpital Yves Le Foll, Saint-Brieuc
  - Site 14, Toulon
  - Site 11, Villefranche-sur-Saône

REFERENCES:
- [Derived] Auliac JB, Fournier C, Audigier Valette C, Perol M, Bizieux A, Vinas F, Decroisette Phan van Ho C, Bota Ouchlif S, Corre R, Le Garff G, Fournel P, Baize N, Lamy R, Vergnenegre A, Arpin D, Marin B, Chouaid C, Gervais R. Impact of Continuing First-Line EGFR Tyrosine Kinase Inhibitor Therapy Beyond RECIST Disease Progression in Patients with Advanced EGFR-Mutated Non-Small-Cell Lung Cancer (NSCLC): Retrospective GFPC 04-13 Study. Target Oncol. 2016 Apr;11(2):167-74. doi: 10.1007/s11523-015-0387-4. PMID 26315967